CLINICAL TRIAL: NCT02267538
Title: Impact of Dexmedetomidine on the Incidence of Postoperative Delirium in Patients After Cardiac Surgery: a Randomized, Double-blinded, and Placebo-controlled Clinical Trial
Brief Title: Dexmedetomidine and Delirium in Patients After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PekingUFH
Record Dates: First submitted 2014-10-09; First posted 2014-10-17 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Delirium; C.Surgical Procedure; Cardiac; Postoperative Complications
Keywords: Delirium; Cardiac Surgical Procedures; Postoperative Complications; Dexmedetomidine; Prevention
MeSH Terms: conditions — Delirium; Postoperative Complications | interventions — Dexmedetomidine; Injections; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dex group (Experimental): The intervention drug (dexmedetomidine hydrochloride for injection) will be administered during a period from before anesthesia induction until the end of mechanical ventilation after surgery.
  Interventions: Drug: dexmedetomidine hydrochloride for injection
- Placebo group (Placebo Comparator): The placebo drug (normal saline, i.e., 0.9% sodium chloride for injection) will be administered in the same way and rate for a same duration as that in the Dex group.
  Interventions: Drug: 0.9% sodium chloride for injection

INTERVENTIONS:
Drug: dexmedetomidine hydrochloride for injection — Before anesthesia, dexmedetomidine hydrochloride for injection (200 ug/2 ml) will be diluted with normal saline to 50 ml (final dexmedetomidine concentration 4 ug/ml).
  Before the induction of anesthesia, a loading dose will be administered by intravenous infusion at a rate of [0.9*kg] ml/h for 10 minutes (i.e., dexmedetomidine 0.6 μg/kg in 10 minutes), followed by continuous infusion at a rate of [0.1*kg] ml/h (i.e., dexmedetomidine at a rate of 0.4 μg /kg/h) until the end of surgery.
  At the end of surgery, the infusion rate will be decreased to [0.025*kg] ml/h (i.e., dexmedetomidine at a rate of 0.1 ug/kg/h) and continued until the end of mechanical ventilation after surgery.
  Other Names: Aibeining (trade name)
  Arms: Dex group
Drug: 0.9% sodium chloride for injection — Before anesthesia, 0.9% sodium chloride for injection 50 ml will be prepared.
  Before the induction of anesthesia, a loading dose will be administered by intravenous infusion at a rate of [0.9*kg] ml/h for 10 minutes, followed by continuous infusion at a rate of [0.1*kg] ml/h until the end of surgery.
  At the end of surgery, the infusion rate will be decreased to [0.025*kg] ml/h and continued until the end of mechanical ventilation after surgery.
  Other Names: normal saline
  Arms: Placebo group

SUMMARY:
Postoperative delirium (POD) is a frequently occurring complication after cardiac surgery. Its occurrence is associated with worse outcomes of patients, including increased morbidity, prolonged hospital stay, increased medical cost, and higher mortality. It is also associated with long-term cognitive decline and decreased quality of life. However, until recently, pharmacological interventions that can effectively prevent its occurrence are still limited. The purpose of this study is to investigate whether perioperative dexmedetomidine use can decrease the incidence of postoperative delirium in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Delirium is a state of global cerebral dysfunction manifested by acute disturbance of consciousness, attention, cognition and perception. It develops over a short period of time (usually hours to days) and tends to fluctuate during the course of the day. The reported incidences of delirium after cardiac surgery varied from 21% to 47%. The occurrence of postoperative delirium has significant harmful effects on patients' outcomes, including increased morbidity, prolonged hospital stay, increased medical cost, and higher mortality. Its occurrence is also associated with long-term cognitive decline and decreased quality of life.

The exact pathogenesis that lead to the occurrence of POD are still unclear, and possibly involves mechanisms such as inflammation, pain and sleep deprivation after surgery. Furthermore, it has been shown that anesthesia management might also have exerted some effects. Studies found that avoidance of unnecessary deep anesthesia (under the guidance of Bispectral Index monitoring) decreases the incidence of POD. Theoretically, measures that decreases the requirement of anesthetics while maintaining adequate depth of anesthesia and those that alleviates inflammation and improves postoperative analgesia as well as sleep quality will decrease the incidence of POD.

Dexmedetomidine is a highly selective alpha-2 adrenoreceptor agonists that provides anxiolysis, sedation and modest analgesia with minimal respiratory depression. Studies showed that, when used as an adjunctive anesthetics, dexmedetomidine significantly decreases the requirement of opioid analgesics and other sedatives during anesthesia. A recent study of our group found that continuous infusion of low-dose dexmedetomidine (0.2 ug/kg/h) during the first night after surgery significantly improved subjective sleep quality. Two randomized controlled trials found that, when compared with traditional sedatives (midazolam and propofol) and analgesics (such as morphine), use of dexmedetomidine in patients after cardiac surgery is associated with decreased risk of delirium. However, questions still exist as to whether dexmedetomidine prevent delirium or just does not increase its occurrence since traditional sedatives/analgesics themselves increases the risk of delirium. Furthermore, animal experiments showed that dexmedetomidine inhibits the degree of inflammation induced by endotoxins.

The investigators hypothesize that use of dexmedetomidine as an adjunctive agent during the perioperative period can decrease the incidence of postoperative delirium in patients undergoing cardiac surgery, possibly by decreasing the requirement of anesthetics during surgery, by ameliorating analgesia as well as sleep quality after surgery, and by alleviating the degree of perioperative inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

Patients of 60 years or older who are planning to receive cardiac surgery (CABG and/or valve replacement surgery)

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Refuse to participate;
2. Preoperative history of schizophrenia, epilepsia, Parkinson syndrome, or severe dementia;
3. Inability to communicate in the preoperative period because of severe visual/auditory dysfunction or language barrier;
4. History of brain injury or neurosurgery;
5. Preoperative sick sinus syndrome, severe bradycardia (HR < 50 bpm), second-degree or above atrioventricular block without pacemaker;
6. Severe hepatic dysfunction (Child-Pugh class C);
7. Severe renal dysfunction (requirement of renal replacement therapy);
8. Other conditions that are considered unsuitable for participation.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request.

REFERENCES:
- [Background] Guenther U, Radtke FM. Delirium in the postanaesthesia period. Curr Opin Anaesthesiol. 2011 Dec;24(6):670-5. doi: 10.1097/ACO.0b013e32834c7b44. PMID 21971396
- [Background] Morandi A, Pandharipande PP, Jackson JC, Bellelli G, Trabucchi M, Ely EW. Understanding terminology of delirium and long-term cognitive impairment in critically ill patients. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):267-76. doi: 10.1016/j.bpa.2012.08.001. PMID 23040280
- [Background] Groen JA, Banayan D, Gupta S, Xu S, Bhalerao S. Treatment of delirium following cardiac surgery. J Card Surg. 2012 Sep;27(5):589-93. doi: 10.1111/j.1540-8191.2012.01508.x. PMID 22978835
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Hopkins RO, Jackson JC. Short- and long-term cognitive outcomes in intensive care unit survivors. Clin Chest Med. 2009 Mar;30(1):143-53, ix. doi: 10.1016/j.ccm.2008.11.001. PMID 19186286
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] MacLullich AM, Beaglehole A, Hall RJ, Meagher DJ. Delirium and long-term cognitive impairment. Int Rev Psychiatry. 2009 Feb;21(1):30-42. doi: 10.1080/09540260802675031. PMID 19219711
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Lin SM, Liu CY, Wang CH, Lin HC, Huang CD, Huang PY, Fang YF, Shieh MH, Kuo HP. The impact of delirium on the survival of mechanically ventilated patients. Crit Care Med. 2004 Nov;32(11):2254-9. doi: 10.1097/01.ccm.0000145587.16421.bb. PMID 15640638
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Krenk L, Rasmussen LS. Postoperative delirium and postoperative cognitive dysfunction in the elderly - what are the differences? Minerva Anestesiol. 2011 Jul;77(7):742-9. PMID 21709661
- [Background] Goto T, Maekawa K. Cerebral dysfunction after coronary artery bypass surgery. J Anesth. 2014 Apr;28(2):242-8. doi: 10.1007/s00540-013-1699-0. Epub 2013 Aug 24. PMID 23982856
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Culley DJ, Baxter M, Yukhananov R, Crosby G. The memory effects of general anesthesia persist for weeks in young and aged rats. Anesth Analg. 2003 Apr;96(4):1004-1009. doi: 10.1213/01.ANE.0000052712.67573.12. PMID 12651650
- [Background] Culley DJ, Baxter MG, Yukhananov R, Crosby G. Long-term impairment of acquisition of a spatial memory task following isoflurane-nitrous oxide anesthesia in rats. Anesthesiology. 2004 Feb;100(2):309-14. doi: 10.1097/00000542-200402000-00020. PMID 14739805
- [Background] Bianchi SL, Tran T, Liu C, Lin S, Li Y, Keller JM, Eckenhoff RG, Eckenhoff MF. Brain and behavior changes in 12-month-old Tg2576 and nontransgenic mice exposed to anesthetics. Neurobiol Aging. 2008 Jul;29(7):1002-10. doi: 10.1016/j.neurobiolaging.2007.02.009. Epub 2007 Mar 7. PMID 17346857
- [Background] Wan Y, Xu J, Ma D, Zeng Y, Cibelli M, Maze M. Postoperative impairment of cognitive function in rats: a possible role for cytokine-mediated inflammation in the hippocampus. Anesthesiology. 2007 Mar;106(3):436-43. doi: 10.1097/00000542-200703000-00007. PMID 17325501
- [Background] Baranov D, Bickler PE, Crosby GJ, Culley DJ, Eckenhoff MF, Eckenhoff RG, Hogan KJ, Jevtovic-Todorovic V, Palotas A, Perouansky M, Planel E, Silverstein JH, Wei H, Whittington RA, Xie Z, Zuo Z; First International Workshop on Anesthetics and Alzheimer's Disease. Consensus statement: First International Workshop on Anesthetics and Alzheimer's disease. Anesth Analg. 2009 May;108(5):1627-30. doi: 10.1213/ane.0b013e318199dc72. PMID 19372347
- [Background] Tang J, Eckenhoff MF, Eckenhoff RG. Anesthesia and the old brain. Anesth Analg. 2010 Feb 1;110(2):421-6. doi: 10.1213/ANE.0b013e3181b80939. Epub 2009 Oct 9. PMID 19820235
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Burkhart CS, Dell-Kuster S, Gamberini M, Moeckli A, Grapow M, Filipovic M, Seeberger MD, Monsch AU, Strebel SP, Steiner LA. Modifiable and nonmodifiable risk factors for postoperative delirium after cardiac surgery with cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2010 Aug;24(4):555-9. doi: 10.1053/j.jvca.2010.01.003. Epub 2010 Mar 15. PMID 20227891
- [Background] Abdel-Meguid ME. Dexmedetomidine as anesthetic adjunct for fast tracking and pain control in off-pump coronary artery bypass. Saudi J Anaesth. 2013 Jan;7(1):6-8. doi: 10.4103/1658-354X.109557. PMID 23717223
- [Background] Gerresheim G, Schwemmer U. [Dexmedetomidine]. Anaesthesist. 2013 Aug;62(8):661-74. doi: 10.1007/s00101-013-2206-6. German. PMID 23917892
- [Background] Jalonen J, Hynynen M, Kuitunen A, Heikkila H, Perttila J, Salmenpera M, Valtonen M, Aantaa R, Kallio A. Dexmedetomidine as an anesthetic adjunct in coronary artery bypass grafting. Anesthesiology. 1997 Feb;86(2):331-45. doi: 10.1097/00000542-199702000-00009. PMID 9054252
- [Background] Khalil MA, Abdel Azeem MS. The impact of dexmedetomidine infusion in sparing morphine consumption in off-pump coronary artery bypass grafting. Semin Cardiothorac Vasc Anesth. 2013 Mar;17(1):66-71. doi: 10.1177/1089253212463969. Epub 2012 Oct 29. PMID 23108415
- [Background] Taniguchi T, Kidani Y, Kanakura H, Takemoto Y, Yamamoto K. Effects of dexmedetomidine on mortality rate and inflammatory responses to endotoxin-induced shock in rats. Crit Care Med. 2004 Jun;32(6):1322-6. doi: 10.1097/01.ccm.0000128579.84228.2a. PMID 15187514
- [Background] Xu L, Bao H, Si Y, Wang X. Effects of dexmedetomidine on early and late cytokines during polymicrobial sepsis in mice. Inflamm Res. 2013 May;62(5):507-14. doi: 10.1007/s00011-013-0604-5. Epub 2013 Mar 5. PMID 23463181
- [Background] Can M, Gul S, Bektas S, Hanci V, Acikgoz S. Effects of dexmedetomidine or methylprednisolone on inflammatory responses in spinal cord injury. Acta Anaesthesiol Scand. 2009 Sep;53(8):1068-72. doi: 10.1111/j.1399-6576.2009.02019.x. Epub 2009 Jun 10. PMID 19519725
- [Background] Xiang H, Hu B, Li Z, Li J. Dexmedetomidine controls systemic cytokine levels through the cholinergic anti-inflammatory pathway. Inflammation. 2014 Oct;37(5):1763-70. doi: 10.1007/s10753-014-9906-1. PMID 24803295
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Hempelmann FW. [Protein binding of xipamide (4-chloro-5-sulfamoyl-2',6'-salicyloxylidide]. Arzneimittelforschung. 1975 Feb;25(2):258-9. No abstract available. German. PMID 1173044
- [Background] Guenther U, Popp J, Koecher L, Muders T, Wrigge H, Ely EW, Putensen C. Validity and reliability of the CAM-ICU Flowsheet to diagnose delirium in surgical ICU patients. J Crit Care. 2010 Mar;25(1):144-51. doi: 10.1016/j.jcrc.2009.08.005. Epub 2009 Oct 13. PMID 19828283
- [Background] Luetz A, Heymann A, Radtke FM, Chenitir C, Neuhaus U, Nachtigall I, von Dossow V, Marz S, Eggers V, Heinz A, Wernecke KD, Spies CD. Different assessment tools for intensive care unit delirium: which score to use? Crit Care Med. 2010 Feb;38(2):409-18. doi: 10.1097/CCM.0b013e3181cabb42. PMID 20029345
- [Background] Ritmala-Castren M, Lakanmaa RL, Virtanen I, Leino-Kilpi H. Evaluating adult patients' sleep: an integrative literature review in critical care. Scand J Caring Sci. 2014 Sep;28(3):435-48. doi: 10.1111/scs.12072. Epub 2013 Aug 26. PMID 23980579
- [Background] Gerlach AT, Murphy CV. Dexmedetomidine-associated bradycardia progressing to pulseless electrical activity: case report and review of the literature. Pharmacotherapy. 2009 Dec;29(12):1492. doi: 10.1592/phco.29.12.1492. PMID 19947809
- [Background] Sichrovsky TC, Mittal S, Steinberg JS. Dexmedetomidine sedation leading to refractory cardiogenic shock. Anesth Analg. 2008 Jun;106(6):1784-6. doi: 10.1213/ane.0b013e318172fafc. PMID 18499610
- [Background] Fischer GW, Silverstein JH. Dexmedetomidine and refractory cardiogenic shock. Anesth Analg. 2009 Jan;108(1):380. doi: 10.1213/ane.0b013e31818c0d98. No abstract available. PMID 19095884
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Mu DL, Wang DX, Li LH, Shan GJ, Li J, Yu QJ, Shi CX. High serum cortisol level is associated with increased risk of delirium after coronary artery bypass graft surgery: a prospective cohort study. Crit Care. 2010;14(6):R238. doi: 10.1186/cc9393. Epub 2010 Dec 30. PMID 21192800
- [Background] Verburg AF, Tjon-A-Tsien MR, Verstappen WH, Beusmans GH, Wiersma T, Burgers JS. [Summary of the 'Stroke' guideline of the Dutch College of General Practitioners' (NHG)]. Ned Tijdschr Geneeskd. 2014;158(1):A7022. Dutch. PMID 24397973
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Gorostidi M, Santamaria R, Alcazar R, Fernandez-Fresnedo G, Galceran JM, Goicoechea M, Oliveras A, Portoles J, Rubio E, Segura J, Aranda P, de Francisco AL, Del Pino MD, Fernandez-Vega F, Gorriz JL, Luno J, Marin R, Martinez I, Martinez-Castelao A, Orte LM, Quereda C, Rodriguez-Perez JC, Rodriguez M, Ruilope LM. Spanish Society of Nephrology document on KDIGO guidelines for the assessment and treatment of chronic kidney disease. Nefrologia. 2014 May 21;34(3):302-16. doi: 10.3265/Nefrologia.pre2014.Feb.12464. Epub 2014 Mar 6. English, Spanish. PMID 24798565
- [Background] Jones AE, Puskarich MA. The Surviving Sepsis Campaign guidelines 2012: update for emergency physicians. Ann Emerg Med. 2014 Jan;63(1):35-47. doi: 10.1016/j.annemergmed.2013.08.004. Epub 2013 Sep 23. PMID 24067755
- [Background] Lin YY, He B, Chen J, Wang ZN. Can dexmedetomidine be a safe and efficacious sedative agent in post-cardiac surgery patients? a meta-analysis. Crit Care. 2012 Sep 27;16(5):R169. doi: 10.1186/cc11646. PMID 23016926
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Derived] Li X, Yang J, Nie XL, Zhang Y, Li XY, Li LH, Wang DX, Ma D. Impact of dexmedetomidine on the incidence of delirium in elderly patients after cardiac surgery: A randomized controlled trial. PLoS One. 2017 Feb 9;12(2):e0170757. doi: 10.1371/journal.pone.0170757. eCollection 2017. PMID 28182690
- See also: Different versions of Confusion Assessemnt Method for the Intensive Care Unit (CAM-ICU) and their validation papers were found in this web. — http://www.icudelirium.org/delirium/languages.html

RESULTS

PARTICIPANT FLOW:
Groups:
- DEX Group: participant who received dexmedetomidine
- CTRL Group: participants who recieved normal saline
Period: Overall Study
Arm/Group | DEX Group | CTRL Group
Started | 142 | 143
Completed | 142 | 143
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DEX Group | CTRL Group | Total
Number analyzed (Participants) | 142 | 143 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (5.4) | 67.5 (5.3) | 66.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 95 | 102 | 197
Body Mass Index "kg/m^2" [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (3.4) | 24.9 (2.8) | 25.1 (3.1)
Education (year) [Median (Inter-Quartile Range); unit: years] | 9 [5 to 12] | 9 [5 to 10] | 9 [5 to 12]
Hypertension [Count of Participants; unit: Participants] | 89 | 91 | 180
Arrhythmia [Count of Participants; unit: Participants] | 32 | 29 | 61
Stroke [Count of Participants; unit: Participants] | 26 | 33 | 59
Chronic Obstructive Ppulmonary Disease [Count of Participants; unit: Participants] | 7 | 4 | 11
Diabetes Mellitus [Count of Participants; unit: Participants] | 43 | 49 | 92
Hyperlipidemia [Count of Participants; unit: Participants] | 38 | 61 | 99
Chronic kidney disease [Count of Participants; unit: Participants] | 1 | 7 | 8
Tumor [Count of Participants; unit: Participants] | 7 | 3 | 10
Thyroid disease [Count of Participants; unit: Participants] | 4 | 3 | 7
Smoking [Count of Participants; unit: Participants] | 51 | 66 | 117
Acute myocardial infarction [Count of Participants; unit: Participants] | 17 | 11 | 28
Calcium Channel Blocker [Count of Participants; unit: Participants] | 33 | 45 | 78
Angiotensin Converting Enzyme Inhibitors/Angiotensin Receptor Blockers [Count of Participants; unit: Participants] | 50 | 46 | 96
β-blocker [Count of Participants; unit: Participants] | 63 | 66 | 129
Statins [Count of Participants; unit: Participants] | 63 | 75 | 138
Antiplatelet drugs [Count of Participants; unit: Participants] | 85 | 82 | 167
European System for Cardiac Operative Risk Evaluation [Median (Inter-Quartile Range); unit: units on a scale] — European System for Cardiac Operative Risk Evaluation is a risk model which allows the calculation of the risk of death after a heart operation.
  The model asks for 17 items of information about the patient, the state of the heart and the proposed operation,and uses logistic regression to calculate the risk of death.
  The minimum score is 0 indicating the lowest risk of death after sugery while the maximum score is 35 indicating the highest risk of death after the heart operation
  units on a scale | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]
History of surgery [Count of Participants; unit: Participants] | 55 | 52 | 107
History of general anesthesia [Count of Participants; unit: Participants] | 24 | 24 | 48
New York Heart Association (NYHA) Functional Classification [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It has four categories based on the degree of limitation during physical activity,the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  From Class I to Class IV, the degree of heart failure is increased with more severe symptoms, for example, no shortness of breath when walking, climbing stairs occurs in patient of Class I while symptoms even exist while at rest in patient of Class IV. Population: 28 participants (17 in the DEX group and 11 in the CTRL group) are acute myocardial infarction ,so their cardiac funcion can not be judged by the NYHA function class
  Participants
    number analyzed (Participants) | 125 | 132 | 257
    I | 2 | 2 | 4
    II | 87 | 92 | 179
    III | 33 | 36 | 69
    IV | 3 | 2 | 5
left ventricular ejection fraction (LVEF)% [Median (Inter-Quartile Range); unit: percentage] — Left ventricular ejection fraction (LVEF) is the fraction of blood ejected from Left ventricle with each heart beat,which is calculated by dividing the stroke volume by the end-diastolic volume. In clinical practice, LVEF is most commonly measured by an echocardiogram and serves as a general measure of a person's cardiac function.
  percentage | 64.4 [56.2 to 70.4] | 64.8 [58.2 to 70.6] | 64.7 [57.0 to 70.6]
the American Society of Anesthesiologists (ASA) Classification [Count of Participants; unit: Participants] — The ASA physical status classification system is a system for assessing the fitness of patients before surgery raised by the American Society of Anesthesiologists (ASA).
  The ASA class has 6 levels. From Class 1 to Class 5, the comorbidity of the patient and the risk to surgery operation are both increased. Class 6 is specially scene indicating a brain-dead patient whose organs are being removed for donor purposes.
  Participants
    II | 1 | 2 | 3
    III | 128 | 129 | 257
    IV | 13 | 12 | 25
Mini-Mental State Examination（MMSE）score [Median (Inter-Quartile Range); unit: units on a scale] — The Mini-Mental State Examination (MMSE) is a questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time.
  Administration of the test takes between 5 and 10 minutes and examines functions including registration, attention and calculation, recall, language, ability to follow simple commands and orientation.
  The MMSE scores range from 0 to 30, with higher scores indicating better cognitive function
  units on a scale | 29 [28 to 30] | 29 [28 to 30] | 29 [28 to 30]
Hospital Anxiety and Depression Scale score [Median (Inter-Quartile Range); unit: units on a scale] — Hospital Anxiety and Depression Scale (HADS) is commonly used to determine the levels of anxiety and depression of the patient. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  The HADS scores range from 0 to 42, with higher scores indicating more severe anxiety anddepression.
  units on a scale | 8 [4 to 12] | 8 [4 to 12] | 8 [4 to 12]
Barthe Index(BI)score [Median (Inter-Quartile Range); unit: units on a scale] — The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). It uses ten variables describing ADL and mobility, which index range from 0 to 100, with higher score indicating better daily life activity and a greater likelihood of being able to live at home with a degree of independence following discharge from hospital.
  units on a scale | 100 [95 to 100] | 100 [95 to 100] | 100 [95 to 100]
Delirium [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Delirium
Description: Delirium was assessed with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) twice daily during the first five days after surgery.
Time Frame: During the first five days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 142 | 143
Participants | 7 | 11
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.341, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.23 to 1.65]

2. Secondary Outcome: Cognitive Function
Description: Cognitive function was assessed with the Mini Mental State Examination (MMSE) at baseline (the day before surgery) and on the sixth day after surgery, and with modified telephone interview for cognitive status (m-TICS) on the 30th day after surgery.
  The introduction of MMSE scale has been explained in the baseline part in the result section.
  The Telephone Interview for Cognitive Status-modified scale(m-TICS) is one of the most popular telephone interview-based screening instruments for mild cognitive impairment and dementia. It consists 11 items including wordlist memory, orientation, attention, repetition, conceptual knowledge and nonverbal praxis, which score ranges from 0 to 48, with higher scores indicating better cognitive function
Time Frame: on the sixth day after surgery, and on the 30th day after surgery
Population: 5 patients (3 in CTRL group and 2 in DEX group) did not complete the MMSE test on postoperative day 6;17 patients (12 in CTRL group and 5 in DEX group) did not complete the m-TICS test on postoperative day 30
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 140 | 140
units on a scale
  MMSE score on postoperative day 6 | 29 [27 to 30] | 29 [27 to 30]
  m-TICS score on postoperative day 30: number analyzed (Participants) | 137 | 131
  m-TICS score on postoperative day 30 | 34 [32 to 37] | 34 [32 to 36]
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.830, Wilcoxon (Mann-Whitney) — MMSE; Median Difference (Final Values) = 0
Statistical Analysis 2: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.405, Wilcoxon (Mann-Whitney) — m-TICS; Median Difference (Final Values) = 0

3. Secondary Outcome: Incidence of Non-delirium Complications After Surgery
Description: Non-delirium complications was defined as any conditions other than delirium that occurred during the first 30 days after surgery and required therapeutic intervention.Complications listed here were not considered adverse events in this study.
Time Frame: Occurrence of non-delirium complications will be monitored until 30 days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 142 | 143
Participants
  Stroke | 3 | 3
  New onset arrythmia | 42 | 51
  Pulmonary complications | 15 | 27
  Upper gastrointestinal bleeding | 2 | 4
  Surgical bleeding | 3 | 3
  Wound dehiscence or infection | 11 | 7
  Acute kidney injury | 37 | 44
  IABP assistance | 6 | 12
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; Incidence of total non-delirium complications within 30 days after surgery; Test type: Other; p = 0.214, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.47 to 1.19]
Statistical Analysis 2: Comparison: DEX Group vs CTRL Group; Incidence of stroke within 30 days after surgery; Test type: Other — stroke; p = 0.993, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.20 to 5.08]
Statistical Analysis 3: Comparison: DEX Group vs CTRL Group; Test type: Other — New onset arrythmia; p = 0.274, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.46 to 1.25]
Statistical Analysis 4: Comparison: DEX Group vs CTRL Group; Test type: Other — Pulmonary complications; p = 0.050, Regression, Logistic; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.26 to 1.00]
Statistical Analysis 5: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.423, Regression, Logistic — Upper gastrointestinal bleeding; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.09 to 2.75]
Statistical Analysis 6: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.993, Regression, Logistic — Surgical bleeding; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.20 to 5.08]
Statistical Analysis 7: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.326, Regression, Logistic — Wound dehiscence or infection; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.61 to 4.34]
Statistical Analysis 8: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.378, Regression, Logistic — Acute kidney injur; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.47 to 1.33]
Statistical Analysis 9: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.156, Regression, Logistic — IABP assistance; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.18 to 1.32]

4. Other Pre Specified Outcome: Pain Intensity
Description: Pain intensity was assessed daily at 8 am during the first five days after surgery with the Numeric Rating Scale (NRS, 0 = no pain, 10 = the worst possible pain).
Time Frame: During the first five days after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 142 | 143
units on a scale
  Pain score after surgery(d1), at rest | 3 [1 to 5] | 3 [2 to 5]
  Pain score after surgery(d2), at rest | 4 [2 to 5] | 3 [2 to 5]
  Pain score after surgery(d3), at rest | 3 [2 to 4] | 2 [2 to 4]
  Pain score after surgery(d4), at rest | 2 [1 to 3] | 2 [1 to 3]
  Pain score after surgery(d5), at rest | 2 [1 to 2] | 1 [1 to 2]
  Pain score after surgery(d1), with coughing | 4 [2 to 6] | 4 [3 to 6]
  Pain score after surgery(d2), with coughing | 5 [3 to 6] | 4 [3 to 6]
  Pain score after surgery(d3), with coughing | 4 [3 to 5] | 4 [2 to 5]
  Pain score after surgery(d4), with coughing | 3 [2 to 4] | 3 [2 to 4]
  Pain score after surgery(d5), with coughing | 2 [2 to 3] | 2 [2 to 3]
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the first row in Outcome 4, i.e., Pain score in Day 1 after surgery, at rest between DEX Group and CTRL group; Test type: Other; p = 0.596, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 2: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the second row in Outcome 4, i.e., Pain score in Day 2 after surgery, at rest between DEX Group and CTRL group; Test type: Other; p = 0.743, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 3: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the third row in Outcome 4, i.e., Pain score in Day 3 after surgery, at rest between DEX Group and CTRL group; Test type: Other; p = 0.282, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 4: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the fourth row in Outcome 4, i.e., Pain score in Day 4 after surgery, at rest between DEX Group and CTRL group; Test type: Other; p = 0.368, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 5: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the fifth row in Outcome 4, i.e., Pain score in Day 5 after surgery, at rest between DEX Group and CTRL group; Test type: Other; p = 0.397, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 6: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the sixth row in Outcome 4, i.e., Pain score in Day 1 after surgery, with coughing between DEX Group and CTRL group; Test type: Other; p = 0.486, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 7: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the seventh row in Outcome 4, i.e., Pain score in Day 2 after surgery, with coughing between DEX Group and CTRL group; Test type: Other; p = 0.414, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 8: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the eighth row in Outcome 4, i.e., Pain score in Day 3 after surgery, with coughing between DEX Group and CTRL group; Test type: Other; p = 0.187, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 9: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the ninth row in Outcome 4, i.e., Pain score in Day 4 after surgery, with coughing between DEX Group and CTRL group; Test type: Other; p = 0.127, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 10: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the tenth row in Outcome 4, i.e., Pain score in Day 5 after surgery, with coughing between DEX Group and CTRL group; Test type: Other; p = 0.378, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

5. Other Pre Specified Outcome: Subjective Sleep Quality
Description: Subjective sleep quality was assessed daily at 8 am during the first five days after surgery with the Numeric Rating Scale (NRS, 0 = best sleep, 10 = the worst possible sleep).
Time Frame: During the first five days after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 142 | 143
units on a scale
  Subjective sleep quality after surgery(d1), score | 2 [0 to 5] | 2 [0 to 6]
  Subjective sleep quality after surgery(d2), score | 3 [2 to 6] | 3 [2 to 6]
  Subjective sleep quality after surgery(d3), score | 2 [2 to 5] | 2 [2 to 4]
  Subjective sleep quality after surgery(d4), score | 2 [1 to 4] | 2 [0 to 4]
  Subjective sleep quality after surgery(d5), score | 2 [0 to 3] | 2 [0 to 2]
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the first row in Outcome 5, i.e., subjective sleep quality in Day 1 after surgery, between DEX Group and CTRL group; Test type: Other; p = 0.777, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 2: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the second row in Outcome 5, i.e., subjective sleep quality in Day 2 after surgery, between DEX Group and CTRL group; Test type: Other; p = 0.919, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1]
Statistical Analysis 3: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the third row in Outcome 5, i.e., subjective sleep quality in Day 3 after surgery, between DEX Group and CTRL group; Test type: Other; p = 0.835, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 4: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the fourth row in Outcome 5, i.e., subjective sleep quality in Day 4 after surgery, between DEX Group and CTRL group; Test type: Other; p = 0.321, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 5: Comparison: DEX Group vs CTRL Group; this statistical analysis applies to the fifth row in Outcome 5, i.e., subjective sleep quality in Day 5 after surgery, between DEX Group and CTRL group; Test type: Other; p = 0.174, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

6. Other Pre Specified Outcome: Length of Stay in the Intensive Care Unit
Description: Results was presented as median (95% confidence interval).
Time Frame: From end of surgery until discharge from Intensive Care Unit or 30 days after surgery
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 142 | 143
hours | 45.0 [43.5 to 46.5] | 46.0 [44.8 to 47.2]
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.788, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.82 to 1.31]

7. Other Pre Specified Outcome: Length of Stay in Hospital After Surgery
Description: Results was presented as median (95% confidence interval).
Time Frame: From end of surgery until discharge from hospital or 30 days after surgery
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DEX Group | CTRL Group
Number analyzed (Participants) | 142 | 143
days | 9 [8 to 10] | 9 [8 to 10]
Statistical Analysis 1: Comparison: DEX Group vs CTRL Group; Test type: Other; p = 0.826, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.23]

ADVERSE EVENTS:
Time Frame: From the start of study drug infusion until 24 hours after the end of study drug infusion.
Arm/Group | DEX Group | CTRL Group
All-Cause Mortality (participants affected / at risk) | 2/142 | 4/143
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/143
Other Adverse Events (participants affected / at risk) | 38/142 | 40/143
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEX Group (N=142) | CTRL Group (N=143)
Intraoperative Bradycardia (Cardiac disorders) | 21 (21) | 14 (14) — Heart rate < 45 beat per minute or a decrease of more than 30% from baseline (average value in the ward), and lasting for at least 5 minutes
Intraoperative Hypotension (Vascular disorders) | 10 (10) | 10 (10) — a decrease of systolic blood pressure of more than 30% from baseline (average value in the ward) and lasting for at least 15 minutes
Postoperative Bradycardia (Cardiac disorders) | 2 (2) | 6 (6) — Heart rate < 45 beat per minute or a decrease of more than 30% from baseline (average value in the ward), and lasting for at least 5 minutes
Postoperative Hypotension (Vascular disorders) | 5 (5) | 10 (10) — a decrease of systolic blood pressure of more than 30% from baseline (average value in the ward) and lasting for at least 15 minutes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes